CLINICAL TRIAL: NCT00804141
Title: An Open-Label Study to Evaluate the Long-Term Safety of Subcutaneous MOA-728 for Treatment of Opioid-Induced Constipation in Subjects With Nonmalignant Pain
Brief Title: Study Evaluating Long-Term Safety of MOA-728 in Participants With Opioid-Induced Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3200K1-3358
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Constipation
Keywords: treatment for opioid-induced constipation
MeSH Terms: conditions — Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MOA-728 12 mg QD (Experimental): Participants will receive MOA-728 12 milligrams (mg) SC once daily (QD) for 48 weeks. Dosing could be adjusted to an as needed (PRN) basis with a minimum 1 dose per week and maximum 1 dose per day.
  Interventions: Drug: N-methylnaltrexone bromide (MOA-728)

INTERVENTIONS:
Drug: N-methylnaltrexone bromide (MOA-728) — MOA-728 will be administered as per the dose and schedule specified in the arm.
  Other Names: Relistor

SUMMARY:
This study is designed to evaluate the long-term safety and tolerability of the subcutaneous (SC) injection form of N-methylnaltrexone bromide (MOA-728) for the treatment of opioid-induced constipation in participants with nonmalignant pain. The study consists of a 2-week screening period, a 48-week open-label treatment period and a 2 week follow-up period. Participants will need to agree to self-administer SC injections, complete daily diaries, and check-in via a daily telephone call during the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years or older.
* A history of pain of at least 2 months duration before the screening visit due to documented underlying nonmalignant condition.
* A history of constipation due to opioid use during 1 month before the screening visit.

Exclusion Criteria:

* A diagnosis of significant gastrointestinal (GI) disorder such as bowel obstruction, fecal incontinence or rectal prolapse.
* A history of active inflammatory bowel disease, irritable bowel syndrome, or megacolon within 6 months before the screening visit.
* A history of malignancy, other than basal cell or squamous cell skin carcinoma, within 5 years before the screening visit.
* A history of chronic constipation before initiation of opioid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2008-12-03 (Actual); Primary Completion 2010-09-20 (Actual); Study Completion 2010-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (104):
- United States (79):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Laguna Hills, California
  - Pfizer Investigational Site, Los Gatos, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Brandon, Florida
  - Pfizer Investigational Site, Chiefland, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Port Orange, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Avon, Indiana
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, West Des Moines, Iowa
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Hagerstown, Maryland
  - Pfizer Investigational Site, Hollywood, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Brockton, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Bingham Farms, Michigan
  - Pfizer Investigational Site, Chesterfield, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Traverse City, Michigan
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Biloxi, Mississippi
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Elizabeth, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Great Neck, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Centerville, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Levittown, Pennsylvania
  - Pfizer Investigational Site, Yardley, Pennsylvania
  - Pfizer Investigational Site, Cranston, Rhode Island
  - Pfizer Investigational Site, Huntingdon, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Hurst, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Christiansburg, Virginia
  - Pfizer Investigational Site, Bellevue, Washington
- Pfizer Investigational Site, Broadmeadow, New South Wales, Australia
- Canada (17):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Pfizer Investigational Site, Dartmouth, Nova Scotia
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Mirabel, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint Romuald, Quebec
  - Pfizer Investigational Site, Sainte-Foy, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
- Colombia (2):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
- South Korea (3):
  - Pfizer Investigational Site, Suwon, Kyonggi-do
  - Pfizer Investigational Site, Seoul, Seoul/Korea
  - Pfizer Investigational Site, Seoul
- Spain (2):
  - Pfizer Investigational Site, Badalona, Barcelona/Spain
  - Pfizer Investigational Site, Madrid, Madrid/Spain

REFERENCES:
- [Result] Michna E, Blonsky ER, Schulman S, Tzanis E, Manley A, Zhang H, Iyer S, Randazzo B. Subcutaneous methylnaltrexone for treatment of opioid-induced constipation in patients with chronic, nonmalignant pain: a randomized controlled study. J Pain. 2011 May;12(5):554-62. doi: 10.1016/j.jpain.2010.11.008. Epub 2011 Mar 22. PMID 21429809
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3200K1-3358&StudyName=Study%20Evaluating%20Long-Term%20Safety%20Of%20MOA-728%20In%20Subjects%20With%20Opioid-Induced%20Constipation

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1040 participants who met the inclusion/exclusion criteria were assigned to receive treatment and 1034 of these participants received at least 1 dose of study drug.
Groups:
- MOA-728 12 mg QD: Participants received N-methylnaltrexone bromide (MOA-728, MNTX) 12 milligrams (mg) subcutaneously (SC) once daily (QD) for 48 weeks. Dosing could be adjusted to an as needed (PRN) basis with a minimum 1 dose per week and maximum 1 dose per day.
Period: Overall Study
Arm/Group | MOA-728 12 mg QD
Started | 1040
Received at Least 1 Dose of Study Drug | 1034
Completed | 477
Not Completed | 563
Not completed — Adverse Event | 157
Not completed — Death | 4
Not completed — Failed to return | 96
Not completed — Investigator request | 8
Not completed — Protocol Violation | 85
Not completed — Withdrawal by Subject | 131
Not completed — Lack of Efficacy | 46
Not completed — Other than specified | 30
Not completed — Enrolled but not treated | 6

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- MOA-728 12 mg QD: Participants received MOA-728 12 mg SC QD for 48 weeks. Dosing could be adjusted to PRN basis with a minimum 1 dose per week and maximum 1 dose per day.
Arm/Group | MOA-728 12 mg QD
Number analyzed (Participants) | 1034
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.67 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 669
  Male | 365

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Serious adverse events (SAEs) included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as an AE that emerged during the treatment period. Any TEAEs included both treatment-emergent SAEs and non-serious AEs. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to Week 50
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MOA-728 12 mg QD
Number analyzed (Participants) | 1034
Participants
  Any TEAEs | 817
  SAEs | 104

2. Secondary Outcome: Change From Baseline in Weekly Bowel Movement (BM) Rate Through Follow-up
Description: Weekly BM rate was derived as the total number of BMs reported in a month divided by the total number of days with non-missing BM diary information in the same month, then multiplied by 7 to normalize to a weekly rate. If the total number of days with non-missing BM diary information in a given month was less than 10 days, the weekly BM rate for the month was defined as missing. The weekly BM rate at baseline was calculated based on the screening period (Days -14 to -1). If the total number of days with non-missing BM diary information during the screening period was less than 5 days, the weekly BM rate at baseline was defined as missing.
Time Frame: Baseline, follow-up (14 days [Week 49 to 50])
Population: All participants who received at least one dose of study drug. Here, 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: BM/week
Arm/Group | MOA-728 12 mg QD
Number analyzed (Participants) | 1034
BM/week
  Baseline | 3.9 (2.8)
  Change during follow-up: number analyzed (Participants) | 529
  Change during follow-up | 0.5 (2.7)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 50
Description: All participants who received at least one dose of study drug.
Arm/Group | MOA-728 12 mg QD
Serious Adverse Events (participants affected / at risk) | 104/1034
Other Adverse Events (participants affected / at risk) | 564/1034
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MOA-728 12 mg QD (N=1034)
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 3
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 4
Prinzmetal angina (Cardiac disorders) | 1
Choroiditis (Eye disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Faecal incontinence (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lumbar hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oesophageal achalasia (Gastrointestinal disorders) | 1
Oesophageal dilatation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abasia (General disorders) | 1
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Device dislocation (General disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Sudden death (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Gallbladder disorder (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Polyarteritis nodosa (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Perihepatic abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1
Blood potassium decreased (Investigations) | 1
Nuclear magnetic resonance imaging abnormal (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Head discomfort (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 4
Migraine (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 2
Radiculopathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3
Alcohol abuse (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Intentional drug misuse (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 2
Mental status changes (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1/669 — This is a gender-specific AE. Only female participants were at risk.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Granuloma skin (Skin and subcutaneous tissue disorders) | 1
Shoulder arthroplasty (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOA-728 12 mg QD (N=1034)
Abdominal pain (Gastrointestinal disorders) | 248
Abdominal pain upper (Gastrointestinal disorders) | 69
Diarrhoea (Gastrointestinal disorders) | 171
Nausea (Gastrointestinal disorders) | 158
Flatulence (Gastrointestinal disorders) | 57
Vomiting (Gastrointestinal disorders) | 77
Influenza (Infections and infestations) | 64
Sinusitis (Infections and infestations) | 56
Upper respiratory tract infection (Infections and infestations) | 61
Back pain (Musculoskeletal and connective tissue disorders) | 65
Headache (Nervous system disorders) | 60
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.